CLINICAL TRIAL: NCT00836420
Title: Cerebral Microdialysis in Patients With Fulminant Hepatic Failure
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Dr. Fin Stolze Larsen, consultant, Rigshospitalet, Denmark
Other Study IDs: KF 00/002
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Fulminant Hepatic Failure
Keywords: ammonia; acute liver failure; brain edema; oxidative metabolism; intracranial pressure
MeSH Terms: conditions — Liver Failure, Acute; Brain Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — microdialysate from the brain as part of rutine monitoring
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- liver: patients with acute liver failure
  Interventions: Procedure: no intervention

INTERVENTIONS:
Procedure: no intervention — the value of the clinical use of microdialysis monitoring of the brain

SUMMARY:
Patients with fulminant hepatic failure (FHF) often develop cerebral edema, high intracranial pressure (ICP)that may result in fatal brain damage. The aim in this protocol is to determine if a rise in the brain concentration of glutamate, lactate and pyruvate are involved in development of surges of high ICP in patients with FHF. The study is observatory in nature and also record the influence of any intervention that may e instituted during the course of the critical illness.

DETAILED DESCRIPTION:
Fulminant hepatic failure (FHF) is often complicated by cerebral edema, high intracranial pressure (ICP) and brain death. Accordingly the intracranial pressure is often monitored in such patients in order to be able to institute treatment before high ICP evolves. As routinely done in patients with severe head injury a microdialysis monitoring catheter is also placed under this procedure to measure metabolic changes that are responsible for surges of high ICP. The aim in this descriptive protocol is to determine if a rise in glutamate, lactate and pyruvate concentration in the brain cortex are involved in development of surges of high ICP in patients with FHF. The study is observatory in nature and also record the influence of any intervention during the course of the critical illness.

ELIGIBILITY:
Inclusion Criteria:

* All patients with fulminant hepatic failure

Exclusion Criteria:

* Age below 18 years
* Pregnancy
* Not obtained informed consent
* Suspicion of cancer disease
* No pupil reaction to light

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients with fulminant hepatic failure
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2000-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Brain lactate concentration and intracranial hypertension | 2013
  to determine if brain oxidative metabolism correlates with brain edema and high intracranial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Fin Stolze Larsen, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet Dept Hepatology A-2121, Copenhagen, Denmark

REFERENCES:
- [Background] Tofteng F, Jorgensen L, Hansen BA, Ott P, Kondrup J, Larsen FS. Cerebral microdialysis in patients with fulminant hepatic failure. Hepatology. 2002 Dec;36(6):1333-40. doi: 10.1053/jhep.2002.36944. PMID 12447856
- [Background] Bjerring PN, Hauerberg J, Jorgensen L, Frederiksen HJ, Tofteng F, Hansen BA, Larsen FS. Brain hypoxanthine concentration correlates to lactate/pyruvate ratio but not intracranial pressure in patients with acute liver failure. J Hepatol. 2010 Dec;53(6):1054-8. doi: 10.1016/j.jhep.2010.05.032. Epub 2010 Aug 3. PMID 20800925
- [Background] Bjerring PN, Hauerberg J, Frederiksen HJ, Jorgensen L, Hansen BA, Tofteng F, Larsen FS. Cerebral glutamine concentration and lactate-pyruvate ratio in patients with acute liver failure. Neurocrit Care. 2008;9(1):3-7. doi: 10.1007/s12028-008-9060-4. PMID 18250976
- [Background] Tofteng F, Hauerberg J, Hansen BA, Pedersen CB, Jorgensen L, Larsen FS. Persistent arterial hyperammonemia increases the concentration of glutamine and alanine in the brain and correlates with intracranial pressure in patients with fulminant hepatic failure. J Cereb Blood Flow Metab. 2006 Jan;26(1):21-7. doi: 10.1038/sj.jcbfm.9600168. PMID 15959460